CLINICAL TRIAL: NCT05315687
Title: Safety and Efficacy of Radioembolization of Metastatic Breast Cancer to the Liver as a 2nd/3rd Line Therapy
Brief Title: Radioembolization of Metastatic Breast Cancer to the Liver as a 2nd/3rd Line Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is being closed because PI left Emory
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Sirtex Medical (Industry)
Responsible Party: Principal Investigator, Nima Kokabi, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002373; NCI-2021-03144 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00002373; RAD5251-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-03-22; First posted 2022-04-07 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Carcinoma in the Liver; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (systemic therapy, Y90 radioembolization) (Experimental): Patients receive systemic therapy. Beginning 1-6 weeks after starting systemic therapy, patients also undergo Y90 radioembolization.
  Interventions: Device: Y-90 SIR-Spheres; Procedure: Yttrium-90 Microsphere Radioembolization; Other: Systemic Therapy
- Arm II (systemic therapy) (Active Comparator): Patients receive systemic therapy.
  Interventions: Other: Systemic Therapy

INTERVENTIONS:
Device: Y-90 SIR-Spheres — Y-90 SIR-Spheres
  Arms: Arm I (systemic therapy, Y90 radioembolization)
Procedure: Yttrium-90 Microsphere Radioembolization — Undergo Y90 radioembolization
  Other Names: Yttrium Y 90 Microsphere Therapy; Yttrium-90 Radioembolization
  Arms: Arm I (systemic therapy, Y90 radioembolization)
Other: Systemic Therapy — Systemic Therapy

SUMMARY:
This phase II trial studies the effects of radioembolization with yttrium Y-90 works as a 2nd or 3rd line therapy for treating patients with breast cancer that has spread to the liver (metastatic to the liver). Yttrium Y-90 radioembolization is a therapy that injects radioactive particles directly into an artery that feeds liver tumors to cut off their blood supply.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of Y90 radioembolization as a 2nd or 3rd line therapeutic option in conjunction with systemic therapy by assessing progression free survival (PFS).

SECONDARY OBJECTIVES:

I. To evaluate the safety of Y90 radioembolization as a 2nd or 3rd line therapeutic option in conjunction with systemic therapy by evaluating treatment related toxicities and identifying baseline predictors of treatment related toxicity.

II. To evaluate the impact of tumor biology i.e. triple negative breast cancer (TNBC) versus (vs.) non-TNBC on PFS and toxicity.

III. To evaluate quality of life (QOL) changes in patients receiving Y90 versus others.

IV. To evaluate the survival (OS) benefit of addition of Y90 radioembolization to systemic therapy.

V. To evaluate compare inflammatory changes in the in the targeted tumors before and after Y90 radioembolization for identification of potential synergistic immunotherapy pathways.

VI. To identify genetic biomarkers of treatment response to Y90 radioembolization.

VII. Evaluation of efficacy and accuracy of hepatobiliary iminodiacetic acid (HIDA) scan as a tool to objectively quantify baseline and post treatment hepatic dysfunction.

VIII. Evaluating timing of Y90 relative to lines of therapies already utilized and disease course.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive systemic therapy. Beginning 1-6 weeks after starting systemic therapy, patients also undergo Y90 radioembolization.

ARM II: Patients receive systemic therapy.

After completion of study treatment, patients are followed up at 4-8 weeks, and then every 12-16 weeks for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Biopsy proven metastatic breast cancer to the liver (liver biopsy including routine genetic profiling) if not performed before, the biopsy will be performed at the time of shunt of study/mapping.
* The metastatic breast cancer to the liver or the primary metastatic breast cancer with one of the following receptor profiling: 1. Triple Negative Breast Cancer (TNBC) (i.e ER-, PR-, HER2-); 2. ER+, PR+, HER2-; 3. ER+, PR-, HER2-; 4. ER-, PR+, HER2-. HER2 negative breast cancer is defined as IHC result of 0 or 1+ in a core needle biopsy specimen of primary breast cancer.
* Tumor burden =< 50% of liver
* Baseline HIDA scan demonstrating normal liver function
* No radiographic, clinical or biopsy evidence of cirrhosis
* Patients to be enrolled in either arm of the study should be deemed appropriate candidate for permissible lines of systemic therapies
* If applicable, patients must have stable brain metastasis (mets) defined as unchanged CNS disease in the past 6 months.
* Life expectancy > 12 weeks as determined by the Investigator
* Hemoglobin >= 8.0 g/dl (within 28 days of cycle 1 day 1)
* White blood cell (WBC) >= 1500/uL (after at least 7 days without growth factor support or transfusion) (within 28 days of cycle 1 day 1)
* Absolute neutrophil count (ANC) >= 1,000/mcL (after at least 7 days without growth factor support or transfusion) (within 28 days of cycle 1 day 1)
* Platelets >= 50,000/mcL (no transfusions allowed within 7 days of day 1 to meet entry criteria) (within 28 days of cycle 1 day 1)
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 (within 28 days of cycle 1 day 1)
* Total bilirubin =< 2 X institutional upper limit of normal (ULN) (within 28 days of cycle 1 day 1)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 5X institutional upper limit of normal (ULN) (within 28 days of cycle 1 day 1)
* Serum creatinine =< 2 mg/dL (or glomerular filtration rate >= 40 mL/min) (within 28 days of cycle 1 day 1)
* Lipase and amylase =< 1.5 x ULN (within 28 days of cycle 1 day 1)
* The effects of Y90 radioembolization/chemotherapy on the developing human fetus are unknown. For this reason, female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy
* FCBP and men treated or enrolled on this protocol must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry for the duration of study participation, and X months after completion of treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* A female of childbearing potential (FCBP) is a sexually mature woman who:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months. This will be assess during screening's H&P by reviewing with subject her reproductive history.
* No surgery, radiotherapy, chemotherapy, immunotherapy, or investigational therapy within 14 days of initiation of therapy on study
* Willingness and ability of the subject to comply with scheduled visits, drug & device administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation

Exclusion Criteria:

* HER2+ breast cancer regardless of ER and PR status.
* Patients who have had chemotherapy or within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier (i.e., have residual toxicities > grade 1)
* Patients who are receiving any other investigational agents or an investigational device within 14 days before starting treatment
* Any prior liver directed intervention (surgical or liver directed therapy for metastatic breast cancer)
* Extrahepatic disease (other than permissible criteria described above).
* Patient with insurance denial for Y90 treatment Consented participants for which Y90 treatment pre-certification was not obtained. This subjects will be considered as a screen failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Liver and overall progression free survival (PFS) | From date of randomization to date of progression or death, where those alive without progression are censored at date of last imaging scan, assessed up to 24 months
  Progression of disease is defined objectively by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 using magnetic resonance imaging (MRI) or computed tomography (CT) and/or by positron emission tomography (PET) using PET Response Criteria in Solid Tumors (PERCIST) criteria. PFS will be estimated using the Kaplan-Meier method, and treatment groups will be compared using log-rank tests. Median PFS will be reported, along with a 95% confidence interval estimated using the Brookmeyer-Crowley method.

SECONDARY OUTCOMES:
Liver progression free survival (PFS) | From date of randomization to date of liver progression or death, where those alive without liver progression are censored at date of last imaging scan, assessed up to 24 months
  Liver progression is defined as progression of disease in the liver only by RECIST 1.1 or PERCIST criteria. Liver PFS will be estimated using the Kaplan-Meier method, and treatment groups will be compared using log-rank tests. Median liver PFS will be reported, along with a 95% confidence interval estimated using the Brookmeyer-Crowley method.

CONTACTS AND LOCATIONS:
Overall Officials: Nima Kokabi, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Wu R, Gogineni K, Meisel J, Szabo S, Thirunavu M, Friend S, Bercu Z, Sethi I, Natarajan N, Switchenko J, Levy J, Abdalla E, Weakland L, Kalinsky K, Kokabi N. Study Protocol: Efficacy and Safety of Radioembolization (REM) as an Early Modality (EM) Therapy for Metastatic Breast Cancer (BR) to the Liver with Y90 (REMEMBR Y90). Cardiovasc Intervent Radiol. 2022 Nov;45(11):1725-1734. doi: 10.1007/s00270-022-03254-4. Epub 2022 Aug 25. PMID 36008574